CLINICAL TRIAL: NCT04826939
Title: Validity (and Reliability) of Two Forms of an Accelerometer-Based Intravaginal Device for Detecting Pelvic Floor Motion
Brief Title: Intravaginal Devices for Pelvic Floor Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Renovia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 13114
Record Dates: First submitted 2021-03-04; First posted 2021-04-01 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Device usage (Experimental): All participants will complete a survey and undergo an evaluation to test the movement of their pelvic floor with the PFDx device and leva device
  Interventions: Device: PFDx device and leva device

INTERVENTIONS:
Device: PFDx device and leva device — Participants will use the leva device, PFDx device and undergo ultrasound measurements during pelvic floor motion to compare the three measurements.

SUMMARY:
The leva and PFDx devices accurately reflect pelvic floor motion consistent with TPUS evaluation. During a voluntary PFM contraction, the change in angle from a position of rest to maximal effort that is detected by each device is positively correlated with TPUS measurements and Modified Oxford scores.

DETAILED DESCRIPTION:
Thirty women 18 years or older will be recruited from OB/GYN, FPMRS or other clinics. Following informed consent and successful screening, subjects will undergo testing as outlined below. Five subjects (all will be invited until five subjects have agreed) will return to clinic in 1-2 weeks to undergo repeat testing using all modalities.

After obtaining informed consent, subject information will be collected, including demographic data, BMI, and medical history (including ob/gyn history). Subjects will complete urinalysis for pregnancy. Subjects will also complete the Pelvic Floor Distress Inventory (PFDI-20) questionnaire. All subjects will undergo a complete pelvic examination including pelvic organ prolapse quantification (POP-Q), a digital assessment of PFM strength (Modified Oxford Scale) and receive a TPUS. Subjects will also complete a series of PFM contractions using the leva and PFDx devices to measure angle changes, and undergo vaginal assessment with a perineomter.

Pelvic floor muscle assessment Prior to recording device measurements, a correct pelvic floor muscle contraction will be verified via manual pelvic floor assessment. Subjects will be instructed to perform a "lift-and-squeeze" maneuver of the pelvic floor, and correct PFM contraction will be verified by the primary examiner (LHQ). PFM strength will then be assessed via digital palpation by the examiner inserting the first and/or second fingers approximately 4 cm into the vagina and palpating the right and left PFM during contraction. Strength will be graded according to the 6-point Modified Oxford Scale (0=no contraction; 1='flicker'; 2=weak; 3=moderate; 4=good; 5=strong). The mean score of the right and left sides of the vagina will be calculated and used for correlation analysis.

Perineometry PFM strength will be measured using a Peritron™ perineometer, which is a 28mm diameter compressible probe connected to a handheld microprocessor. It provides readings of pelvic floor contraction in cm of H20 with precision up to one decimal point, and it has been demonstrated to show reproducible and reliable measurements. The resting vaginal pressure and two peak pressures will be measured. For this study, PFM strength is defined as the augmented vaginal pressure, calculated by measuring the average of 2 peak pressures minus the resting vaginal pressure.

TPUS measurements TPUS imaging will be completed at the time of the study visit using the BK Medical Ultrafocus (Peabody, MA) and 8802 transperineal transducer. The probe will be covered with ultrasound gel and a probe cover. All ultrasound studies will be performed in the office setting with the patient in the dorsal lithotomy position, with hips flexed and abducted. No preparation is required, and no rectal or vaginal contrast will be used. Patients will be instructed to arrive at the office with a partially full bladder and to avoid excessive pressure on surrounding structures that might distort the anatomy. In the sagittal view, dynamic ultrasound parameters will be measured relative to a horizontal reference line at the level of the infero-posterior margin of the pubic symphysis. Dynamic images will be obtained during PFM contractions and at rest. At least 3 cycles of PFM contraction and relaxation will be recorded for each individual.

Baseline assessment will be performed at rest, then with 3 maximum-effort voluntary contraction (MVC). Ultrasound measurements will include: Anterior-posterior distance (APD) of the levator hiatus to the pubic bone (primary aim), levator urethra gap (LUG), distance from bladder neck to the pubic bone and distance of the midurethra to the pubic bone. Urethral angle at rest and with max contraction will also be measured. The cravioventral shift of the levator plate relative to a vertical line of reference relative to the anorectal angle will also be measured.

Leva measurements Subjects will be instructed on proper insertion and placement of the leva device. The examiner will assist with device placement, as needed. With the leva inserted, subjects will assume a standing position. Subjects will complete a series of pelvic floor muscle training (five lifts for 15 seconds of maximum lift, followe by 15 seconds of rest).

PFDx measurements The examiner will place the PFDx in the vagina, ensuring the ring component is positioned at the fornix with the extension running the length of vagina and out of the body. With the device retained in the vagina, subjects will assume a standing position. Angle measurements will be recorded at rest and with maximal voluntary 'lift-and-squeeze' contraction. These measurements will be repeated at least 3 times with 1-minute rest between each measurement.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Presence of a vagina
* Ability to read and write English
* BMI <30
* Reports they are able to perform a kegel exercise

Exclusion Criteria:

* Inability to perform a kegel exercise
* Pelvic organ prolapse greater than ICS POP-Q Stage II
* Known, untreated pelvic, vaginal or urinary tract infection
* Currently pregnant

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Validate leva measurements with transperineal ultrasound (TPUS) | Through final study visit (about 3 months)
  During a voluntary pelvic floor muscle contraction, the change in angle from a position of rest to maximal effort that is detected by the leva device will be compared to the change in distance from the pubic bone to the levator plate measured by 2D TPUS during the same task.

SECONDARY OUTCOMES:
Compare leva angle change measurements with Modified Oxford, Brinks | Through final study visit (about 3 months)
  Modified Oxford, Brinks is a commonly used clinical assessment tool to measure pelvic floor muscle strength
Compare PFDx angle change measurements with Modified Oxford, Brinks | Through final study visit (about 3 months)
  Modified Oxford, Brinks is a commonly used clinical assessment tool to measure pelvic floor muscle strength
Compare PFDx to a perineometer | Through final study visit (about 3 months)
  Measuring angle change measurements with change in vaginal squeeze pressure
Compare leva to a perineometer | Through final study visit (about 3 months)
  Measuring angle change measurements with change in vaginal squeeze pressure
Determine the test-retest reliability of Manual muscle testing angle measurements over 2 time points | Through final study visit (about 3 months)
  Time points are 1-2 weeks apart
Determine the test-retest reliability of perineometry angle measurements over 2 time points | Through final study visit (about 3 months)
  Time points are 1-2 weeks apart
Determine the test-retest reliability of ultrasound angle measurements over 2 time points | Through final study visit (about 3 months)
  Time points are 1-2 weeks apart
Determine the test-retest reliability of leva angle measurements over 2 time points | Through final study visit (about 3 months)
  Time points are 1-2 weeks apart
Determine the test-retest reliability of PFDx angle measurements over 2 time points | Through final study visit (about 3 months)
  Time points are 1-2 weeks apart

CONTACTS AND LOCATIONS:
Overall Officials: Lieschen Quiroz, MD, Principal Investigator — University of Oklahoma HSC
Locations (2):
- United States (2):
  - OU Physicians, Oklahoma City, Oklahoma
  - University ofOklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No
No plans to share information